CLINICAL TRIAL: NCT04381416
Title: Pre-pivotal, Randomized Study to Assess the Safety and Efficacy of the IUB SEAD™ Device in Women Suffering From Abnormal Uterine Bleeding
Brief Title: Study to Assess the Safety and Efficacy of the IUB SEAD™ Device
Acronym: AUB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ocon Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 55P112
Record Dates: First submitted 2020-05-04; First posted 2020-05-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Abnormal Uterine Bleeding
MeSH Terms: conditions — Metrorrhagia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort I: SEAD treatment (Experimental): Following the first SEAD™ treatment, women who experience a sub-optimal treatment response (at least 3 months after the first treatment) will be eligible to receive a second SEAD™ treatment (see re-treatment criteria below), which will be performed during the first 1-3 days following the cessation of their menses immediately following decision to retreat.
  Interventions: Device: SEAD treatment
- Cohort II: Repeted SEAD treatment 1m post op (Experimental): Following the first SEAD™ treatment, women will undergo a second SEAD™ treatment during the first 1-3 days following the cessation of their next menses.
  Interventions: Device: SEAD treatment

INTERVENTIONS:
Device: SEAD treatment — up to two 30-min endometrial ablation sessions using the IUB SEAD™ device, in a hospital outpatient clinic

SUMMARY:
Pre-pivotal, randomized study to assess the safety and efficacy of the IUB SEAD™ device in women suffering from abnormal uterine bleeding.

DETAILED DESCRIPTION:
Chronic abnormal uterine bleeding (AUB), involving menstrual bleeding of abnormal quantity, duration, or schedule, is experienced by 10-35% of women, and can markedly impact everyday activities, can lead to iron deficiency and in severe cases, can necessitate emergency medical care.

While pharmacologic treatment options exist, some women desire a treatment that requires less maintenance or is definitive. Endometrial ablation is a minimally invasive approach applied to manage AUB and can be performed using resectoscopic instruments or with a non-resectoscopic approach, in which the device is inserted into the uterine cavity and delivers energy to uniformly destroy the uterine lining. Non-resectoscopic endometrial ablation has become an accepted office-based procedure, but requires training in administration and response to complications of conscious sedation and of assisting personnel.

The IUB SEAD™ device is a novel Spherical Endometrial Ablation Device, developed to allow for a simple, office-based chemical endometrial ablation to treat AUB. The suggested procedure is expected to be simpler than the currently available ablation methods and to result in a clinically meaningful delay or abolishment of the need for hysterectomy

ELIGIBILITY:
Inclusion Criteria:

1. Female subject age 35 to 50 years, inclusive
2. Suffering from heavy menstrual bleeding with no definable organic cause and are candidates for global endometrial ablation or surgical treatment
3. Have a histological finding in a recent (max 4-month-old, with a window of 1 month) endometrial biopsy (Pipelle® or other non-treatment-based biopsy) that demonstrates benign endometrial histology: proliferative endometrium and/or disordered endometrium and/or histological findings associated with dysfunctional endometrium (e.g. irregular shading, un-ovulatory bleeding and such); no histological findings of hyperplasia are allowed
4. Premenopausal status confirmed by FSH level measurement at screening (FSH < 40 IU/L). FSH level measurement will be repeated in case of a borderline result
5. Screening hemoglobin levels >9.0 g/dL
6. Uterine sound measurement of 6.5-11 cm (external os to internal fundus)
7. PBAC score of >150 for 3 months prior to study treatment or PBAC score >150 one month prior to study treatment for women who had at least 3 prior months (documented) of failed medical therapy
8. Predictable, cyclic menstrual cycles
9. Negative serum pregnancy test at the Screening visit and on the day of SEAD™ treatment
10. Sexually active women must agree to use an effective method of contraception throughout the course of the study. For this study, effective methods of contraception are considered to be those listed below:

    * Barrier method, i.e., (a) condom (male or female) with spermicide or (b) diaphragm with spermicide or
    * Vasectomy (partner), or
    * Abstinence, if in line with the preferred and usual lifestyle of the subject [where abstinence is defined as refraining from heterosexual intercourse]
11. Subject able to understand and sign a written informed consent form
12. Subject willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures
13. Demonstrates an understanding of how to record menstrual blood loss using a menstrual pictogram

Exclusion Criteria:

1. Pregnant women or those who desire to conceive at any time in the future
2. Congenital malformation of the uterine cavity (bicornuate, septate)
3. Inability to visualize the uterine cavity because of intracavitary pathology and/or significant uterine asymmetry, including patients with submucous myomas and/or polyps and synechiae that heavily distort the uterine cavity
4. Underwent prior uterine surgery that interrupts the integrity of the uterine wall (e.g., transmural myomectomy, classical Cesarean section, endometrial ablation, hysteroscopic resection) or a uterine biopsy accompanied by curettage in the last 12 months
5. Have abnormal endometrial biopsy (i.e., unresolved adenomatous complex hyperplasia, endometrial cancer)
6. Have a documented clinical history of metal allergy or hypersensitivity
7. Suffers from active endometritis, active pelvic inflammatory disease (PID) or active sexually transmitted disease (STD)
8. Suffers from active infection of the genitals, vagina, cervix, or uterus
9. Presence of bacteremia, sepsis, or other active systemic infection
10. Known/suspected abdominal, pelvic, or gynecological malignancy within the past 5 years
11. Known clotting defects or bleeding disorders or subjects who went through blood transfusion (for any reason) in the three months prior enrollment
12. Currently using anticoagulant treatment
13. Subjects with abnormal Papanicolaou (Pap) test or atypical squamous cells of undetermined significance (ASCUS) with positive high-risk human papilloma virus (HPV) test result within the appropriate screen timeframe, and prior to SEAD™ treatment. Alternatively, a colposcopy performed prior to SEAD™ treatment, that showed evidence of dysplasia requiring treatment. In case treatment was performed > 6 months prior to enrollment and follow-up was done with no evidence of disease by clinical evaluation, the subject is eligible.
14. Previously had endometrial ablation procedure of any kind
15. Suffers from clinically significant adenomyosis indicated by subject complaints, imaging or clinician's judgment
16. Presence of an implantable contraceptive device
17. Post-partum ≤ 6-months
18. Currently participating in or considering participation in a research study of an investigational drug or device that would begin during the course of this investigational study
19. Any general health or mental, or other situation or condition which, in the opinion of the Investigator, could present an increased risk for the subject or impact the subject's ability to comply with protocol requirements.

Ages: 35 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — premenopausal women suffering from AUB
Enrollment: 16 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Adverse events | 12 months
  assess the 12-month safety of IUB SEAD treatment in women suffering from AUB.
Pictorial Blood Loss Assessment Chart changes from baseline | 12 months
  To assess the efficacy of IUB SEAD treatment in women suffering from AUB, 12 months after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Rouemen Velev, Md, Principal Investigator — Sheynovo medical center
Locations (1):
- Sheynovo medical center, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No